CLINICAL TRIAL: NCT06745687
Title: A Prospective, Multi-center, Single-arm Clinical Trial of BCMA/CD3 BsAb in the Treatment of High-risk Smoldering Multiple Myeloma
Brief Title: BCMA/CD3 BsAb in the Treatment of High-risk Smoldering Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024009
Record Dates: First submitted 2024-12-10; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: High Risk Smoldering Multiple Myeloma
Keywords: high risk smoldering multiple myeloma; BCMA/CD3 BiTE; CM-336

STUDY DESIGN:
Intervention Model Description: A single-arm multi-center trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CM-336( BCMA/CD3 bispecific antibody) (Experimental): Patients enrolled in the trial will receive CM336 subcutaneously, which is an BCMA/CD3 bispecific antibody therapy.
  Interventions: Drug: CM336

INTERVENTIONS:
Drug: CM336 — Patients received subcutaneous CM-336 80 mg once weekly in 28-d cycles after two step-up priming doses of 3 mg and 20 mg given on day 1 and day 4 of cycle 1 and cycle2. Then patients will be given 160mg every 2 weeks from cycle 3 to cycle 6. The dosing interval is adjusted according to the evaluation of efficacy every 6 cycles from cycle 7 to cycle 24.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of CM-336, which is a BCMA/CD3 BiTE, in the treatment of high risk smoldering multiple myeloma.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of CM-336, which is a BCMA/CD3 BiTE, in the treatment of high risk smoldering multiple myeloma.

High-risk SMM has a high risk of transforming to MM, and there is no unified treatment plan in clinical practice at present. Studies have proved that early treatment can help prevent end organ damage caused by disease progression and improve patient prognosis. The treatment of high-risk SMM needs to be further explored. BCMA/CD3 BITE in the treatment of RRMM shows a high remission rate and low toxicity and side effects, and it is expected to become a potential treatment choice for high-risk SMM patients

ELIGIBILITY:
Inclusion Criteria:

1. Know and voluntarily sign an informed consent form (ICF).
2. Age ≥18 years.
3. Definite diagnosis of SMM: According to IMWG Criteria 10, the patient must have histologically or cytologically confirmed smoldering multiple myeloma (SMM), including:

   1. Serum M protein ≥3 g /dL and/or BMPCs≥10%(but not more than 60%)
   2. No anemia: hemoglobin ≥10 g /dL
   3. No renal failure: serum creatinine ≥2.0 mg/dL
   4. No hypercalcemia: calcium ≥10.5 mg/dL
   5. dissolving bone lesions without radiographic indications: X-ray, CT, or positron emission tomography (PET)/CT without dissolving bone lesions, with no more than 1 lesion on whole-body MRI (Note: In the investigator's judgment, whole-body CT or PET/CT may replace MRI for patients with contraindications or for whom MRI is not available).
   6. FLC ratio <100 (unless light chain ≤10 mg /dL is involved) Note: Anemia, renal failure and hypercalcemia are allowed if there is evidence that anemia, renal failure, hypercalcemia or bone lesions are not associated with multiple myeloma (MM).
4. High-risk SMM are defined as meeting one or more of the three criteria in the following part: (i) Mayo 2018, (ii) IMWG 2020 and (iii) evolving pattern.

   (i)Mayo 2018
   * M protein > 2 g/dL ② The ratio of affected to unaffected FLC was > 20 ③BMPC > 20% of the 3 items meet any 2 or more

   (ii) IMWG 2020
   * FLC ratio 0-10: 0 points 10-25: 2 points 25-40: 3 points >40: 5 points

     ②M protein (g/dL) 0-1.5: indicates 0 points 1.5-3: 3 points >3: 4 points

     ③BMPC (%) 0-15: 0 points 15-20: 2 points 20-30: 3 points 30-40: 5 points >40: 6 points

     ④FISH * : Yes: 2 points None: 0 points The sum of the four points is greater than or equal to 9 （iii）Progression model
   * Necessary condition: BMPC>10% ② Sufficient conditions: a. Serum M protein >3 g/dL b. IgA type SMM c. Immune paralysis (reduction of two uninvolved homologous immunoglobulins) d. The proportion of free light chain (FLC) in serum that is affected/not affected > 8 (but <100) e.M protein level increased (SMM type increased; Serum M protein level was increased by ≥25% twice in 6 months.

   F.BMPC: 50%-59% g. Abnormal plasma cell immunophenotype (95% + of cloned BMPC) and reduction of one or more uninvolved immunoglobulin types.

   h.≥5% of cells had chromosomal abnormalities (t (4,14) or del 17 p or 1 q acquisition i. Increased circulating plasma cells (PCs>5×106/L or 5%) j. Merri indicates diffuse abnormalities or 1 focal lesion, and/or increased uptake of focal lesion in PET-CT class without underlying osteolytic osteopathy. Meet the necessary conditions, 1 or more sufficient conditions.

   *FISH exceptions are defined as the presence of any of the following: t (4,14), t (14,16), 1 q amplification, del 13 qt, t (4,20)
5. ECOG physical status score ≤2 points.
6. Meeting the following laboratory indicators within 28 days prior to study participation:

   a. neutrophils absolute value (ANC) >1000/ml b. Platelet count (PLC)> 75,000 /ml c. Total bilirubin ≤2 mg/dL d. Glutamic oxalic aminotransferase (AST) <2.5 times the conventional upper limit (ULN) e. Alanine aminotransferase (ALT) <2.5 times the upper limit of normal (ULN) f. Estimated creatinine clearance (CLcr)≥60 mL/min.
7. Non-childbearing women meet the entry requirements; Female patients of childbearing age must have a negative serum (beta-human chorionic gonadotropin) or urine pregnancy test at the time of screening.
8. Men, women of childbearing age, and their partners voluntarily use contraception deemed effective by investigators during treatment and for at least three months after CAR T cell transfusion.
9. Male patients must agree not to donate sperm from the initial screening period until 90 days after the last medication.
10. Patients must be willing and able to complete study procedures and follow-up examinations.

Note: Fertile women are all women who have begun menstruating and are not in late menopause and who have not undergone surgical sterilization (e.g., hysterectomy, bilateral tubal ligation, bilateral oophorectomy). Postmenopause is defined as more than 12 consecutive months of amenorrhea for an unspecified reason. Women who are using mechanical birth control methods such as oral contraceptives or intrauterine devices should be considered fertile. Male subjects (including those who have undergone vasectomy) must consent to the use of condoms during sex with women of childbearing age and must not plan to impregnate the woman during the study drug use period from the date of signing the informed consent form and within 3 months after the last study drug receipt.

Exclusion Criteria:

1. Diagnosis of symptomatic multiple myeloma: refer to the Chinese Guidelines for Diagnosis and Treatment of multiple myeloma (revised in 2022);
2. Along with other tumors that must be treated.
3. Previously received immunotherapy against BCMA targets.
4. The researchers judged that BCMA/CD 3 dual antibody therapy is not suitable, such as severe cardiopulmonary disease and other conditions that are not suitable for BCMA/CD 3 dual antibody therapy.
5. Received SMM treatment within six months.
6. Known intolerance, allergy or contraindications to BCMA/CD 3 dual anti-active ingredients.
7. Patients with unstable or active cardiovascular and cerebrovascular diseases meet any of the following criteria:

   1. Unstable angina pectoris, symptomatic myocardial ischemia, myocardial infarction, or coronary artery reconstruction had occurred within 180 days prior to initial administration.
   2. Uncontrolled hypertension (>140/90 MMHG, with a blood pressure fluctuation of more than 180/100 MMHG over 6 months);
   3. Uncontrolled and clinically significant conduction abnormalities (e.g., patients with ventricular arrhythmias controlled by antiarrhythmic drug therapy), not excluding patients with first-degree AV block or asymptomatic left anterior bundle branch block/right bundle branch block (LAFB/RBBB);
   4. Echocardiographic left ventricular ejection fraction (LVEF) < 40%;
   5. History of stroke or intracranial hemorrhage within 12 months prior to screening;
   6. Severe thrombotic events before treatment.

9) Known active human immunodeficiency virus (HIV) infection or HIV seropositivity.

10) Active hepatitis B or C infection. Screening requires hepatitis serological testing. If hepatitis B surface antigen is positive, a negative DNA polymerase chain reaction (PCR) result is required to be confirmed before enrollment (after anti-HBV treatment, a negative DNA polymerase PCR result is required before enrollment). If the hepatitis C antibody is positive, an RNA PCR test is performed and the result before enrollment is confirmed to be negative.

11) Pregnant or lactating women. 12) Any active gastrointestinal dysfunction that affects the patient's ability to swallow pills, or any active gastrointestinal dysfunction that may affect the absorption of investigational therapeutic drugs.

13) Patients had major surgery (for example, requiring general anesthesia) within 2 weeks before enrollment began, or will not fully recover from surgery, or have surgery scheduled during the time they plan to participate in the study. Kyphoplasty or spondyloplasty is not considered major surgery. Note: Patients who plan to perform surgery under local anesthesia may participate in the study.

14) Received live attenuated vaccine within 4 weeks prior to administration of the first investigational drug.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
minimal residual disease netativity(MRD negativity) | baseline, 28 days per cycle, cycle 6 day 28, cycle 12 day 28, cycle 18 day 28, cycle 24 day 28, 1 year and 2 year after end of treatment.
  The proportion of abnormal plasma cells occupying nuclear cells in the samples
Adverse events and serious adverse events | up to 2 years
  Adverse events (AEs), serious adverse events (SAEs), and assessments of clinical laboratory values

SECONDARY OUTCOMES:
time to response | up to 2 years
  Time from randomization to first documentation of hematologic response
Hematologic response rate | up to 2 years
  Overall hematologic (CR + VGPR + PR) response rate based on central laboratory results based on 2016 IMWG response criteria.
progression free survival(PFS) | up to 2 years after end of therapy
  progression free survival defined as time from randomization to date of hematologic progression or documented disease progression (PD). Patients without documentation of death at the time of analysis were censored at the date last known to be alive
overall survival(OS) | up to 2 years after end of therapy.
  Time from randomization to date of death. Patients without documentation of death at the time of analysis were censored at the date last known to be alive
duration of response(DOR) | up to 2 years after end of therapy
  DOR is defined as the time from initiation of first response to first documentation of disease progression or death whichever occurs first. Patients without documentation progressed or died are censored at the date last known progression-free.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China